CLINICAL TRIAL: NCT00355459
Title: A Prospective Clinical Study Assessing the Effects of Tetracycline Antibiotic on Tear Film and Tear Lipid Composition Within a Population of Patients Diagnosed With Blepharitis and Dry Eye Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has elected to terminate study at this time
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 082005-026
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Dry Eye Syndrome
Keywords: Meibomian Gland Dystrophy
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: Tetracycline: Doxycycline analog

SUMMARY:
The purpose of this research project is to determine the effects of oral tetracycline such as Minocycline (Minocin) on tear film composition and tear lipid (meibomian gland secretions) characteristics in patients with chronic Blepharitis and associated dry eyes.

DETAILED DESCRIPTION:
Tear film dysfunctions, which are collectively diagnosed as dry eye syndromes and Meibomian Gland Dystrophy (MGD) afflict millions of individuals worldwide, more than 10 million in the United States alone. Typically, symptoms include ocular burning, foreign body sensation, photophobia, redness and other symptoms that result in overall chronic discomfort in patients. Tetracycline analogues, such as minocycline, have demonstrated effectiveness in treating primary meibomianitis, one type of chronic blepharitis and have been prescribed to patients for sometime. It has been demonstrated that tetracycline can inhibit lipase activity and therefore decrease the release of noxious free fatty acids. Tetracycline also inhibits bacterial lipase activity in vitro and has other effects. We have been investigating the associations between chronic blepharitis and eyelid meibomian gland lipids and microflora for a number of years and have discovered important relationships between these lipids and chronic blepharitis disease states. Because of its high concentration 12 hours post dose, low renal clearance, long half life, and high level of binding to serum proteins, minocycline has been suggested as a good treatment option. The study proposes to determine the effect of oral treatment with tetracycline analogues on the Tear Film and Tear Lipid Composition within a Population of Patients Diagnosed with Dry Eye Disease and Meibomian Gland Dysfunction.

Patients diagnosed with dry eye syndrome as well as Meibomian Gland Dystrophy (MGD) will be selected to participate in a clinical study: baseline visit, 1-month following initiation of treatment, 3-months after initiation of treatment, and 3-months after discontinuation of treatment.

Once assessed and qualified to take part in the trial, participants will undergo the following tests during each visit:

I. Ocular assessment of signs and symptoms II. Evaporometry III. Fluorophotometery IV. Schirmers Testing V. TBUT VI. Bacteriology VII. Transillumination & Meibography VIII. Meibomian gland expression and lipid analysis

After completion of the baseline visit, each patient will be given a 2-week regimen of 50-mg dose of Minocycline followed by 10-week supply of 100-mg Minocycline to be taken daily after breakfast. In addition, they can continue using artificial tears and additional treatments as prescribed by their treating physicians.

I. Ocular assessment Patients' symptomology as well as the assessors' diagnostic findings will be recorded and reviewed in detail before patient entrance into study. These include visual acuity, biomicroscopy of lids/lashes, conjunctiva, and cornea. Moreover, corneal as well as conjunctival staining will be performed with the use of two colored dyes: Lissamine green and fluorescein. In addition, the investigator will record any pathology with the patients' natural lens, iris, and pupil.

II. Evaporometer: Evaporative flow and contribution to turnover An evaporometer utilizes a pump to direct air through a drying tube (Hammond Drierite, Xenia, OH) into a goggle. The goggle containing a water vapor detector and a temperature monitor is placed firmly over the eye. The pumped air passes into the goggle, reducing the humidity to 15%, at which time the pump is turned off. The increase in humidity due to evaporation from skin or evaporating tears is measured and stored in a computer. The process is carried out first with the eyelids closed and then with them open; the difference is the tear evaporation rate. The area of the interpalpebral ocular surface is used to calculate evaporation per unit area; the image of the area is captured with the use of a digital camera and calculated directly with the aid of computer software (ADOBE Photoshop, version 6.0.1.2001, ADOBE Systems, and San Jose, California). Evaporative outflow as a percentage of available tear volume will be calculated from the rate of the rise of relative humidity inside the goggle with the eye open minus the evaporative contribution of the closed eye skin within the goggle.

The evaporative contribution to turnover will be calculated as evaporative outflow per available tear volume per minute divided by tear turnover.

III. Fluorophotometer: Tear volume, flow and turnover Background fluorescence will be determined prior to the instillation of 0.5 micro liters of 0.5% sodium fluorescein onto the ocular surface. Utilizing a fluorophotometer (Fluorotron Master, Ocumetrics, Mountain View, CA), eight measurements will be taken from each eye to determine tear fluorescence. The first two measurements will be performed one minute apart and subsequent measurements will be repeated with three minute intervals until completion at 19 minutes. This data will be analyzed to calculate tear volume, flow and tear turnover.

IV. Schirmers testing: Quantitative tear measurement performed with and without anesthetic Drops. A commonly used paper wick will be placed between the eyeball and outer third of the lower lid cul-de-sac in order to measure quantitatively the production of tears. This test typically takes 5 minutes to perform.

V. Tear Break-Up Time - Quantitative/Qualitative assessment of corneal and conjunctival dry spots (devitalized surface epithelial cells) A drop of fluorescein will be instilled in both eyes of the patient. Patient will be asked to blink normally for the dye to spread evenly in the eye. Once completed, patient will be asked to blink once and hold eyes open while the assessor uses a stop watch to record number of seconds it takes for the tear film to break-up. This is a tool that allows the examiner to grade the quality of the tear film. Normal control patient TBUT is 10-12 seconds while a dry eye patient TBUT is less than 2 seconds.

VI. Bacteriology - Eyelid microflora evaluation Samples of eyelid and conjunctival microflora of each eye will be taken separately with a calcium alginate swab dipped in 0.9% salt solution. After streaking the swab on different plates (blood agar, chocolate agar, and reduced brucella blood agar), it will placed into a tube of thioglycolate for bacteriological assessment.

VII. Transillumination & Meibography - Quantitative assessment of lower lid meibomian gland lipid production An excretory gland, the primary role of the meibomian glands is to produce and secrete lipids into the tear film. The purpose of this test is to determine quantitatively the number of lower lid glands that are functional lipid producers. A transilluminator (muscle light) with a light dispersing tip will be used to illuminate the glands. The small band of light will transilluminate the inverted lower lids of patients. With the use of a digital camera, a picture will be taken in order to assess vital glands from drop-outs (non-producing glands). This is accomplished with a frame grabber that is matched to a Hitachi KP-F2A progressive scanner infrared camera that is mounted on a slit lamp microscope. Images will be captured and stored with the use of imaging software.

VIII. Meibomian gland expression and lipid analysis - Lower and Upper eye lid samples will be collected and assayed for their biochemical makeup With the use of an ocular conformer and cotton tip applicator, samples of upper and lower lid meibomian gland lipids will be collected and assessed for make-up

ELIGIBILITY:
Inclusion Criteria: Patients over 18 years of age, patient willing and able to comply with the protocol. Insidious onset and greater than three month's duration of ocular symptoms consistent with dry eye and meibomian gland disease. Ocular surface vital staining consistent with aqueous deficient dry eyes with less than +1 conjunctival injection and no more than minimal lid inflammation. Normal controls will also be tested for this trial.

Exclusion Criteria: Any patient with punctual occlusion or punctual plugs within the past 2 months. Patients with active ocular infection or inflammatory disease, history of herpetic keratitis, history of retinal detachment, concurrent contact lens use during the trial period, ocular surgery within the past six months, patients with glaucoma, anterior membrane dystrophy, active trichiasis or any eyelid globe malposition abnormality, e.g., entropion, ectropion, etc. Patients with epiphora (excessive tearing). Moreover, patients taking medications known to effect aqueous tear production or meibomian secretions or use of tetracycline or tetracycline analogs for treatment of other medical conditions within the past 3 months. Patient must not have participated in (or be currently participating in) any investigational therapeutic drug or device trial within the previous 30 days prior to their start date for this trial. In addition, any patient suffering from organic brain syndromes or major psychiatric disorder that would interfere with compliance or subjective reporting will be discouraged from participating in this trial.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Evaporometry
Fluorophotometery
Meibomian gland expression and lipid analysis

SECONDARY OUTCOMES:
Schirmers Testing
TBUT
Bacteriology
Transillumination & Meibography

CONTACTS AND LOCATIONS:
Overall Officials: James P. McCulley, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States